CLINICAL TRIAL: NCT03386500
Title: A Phase 1/2 Trial for Patients With Newly Diagnosed Anal Cancer Treated With Concurrent Radiation Therapy, 5FU, Mitomycin and BMX-001
Brief Title: Safety Study of BMX-001 (Radio-protector) in Patients With Newly Diagnosed Anal Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: BioMimetix JV, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0247-17-FB
Record Dates: First submitted 2017-12-07; First posted 2017-12-29 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-06

CONDITIONS: Anal Cancer, Squamous Cell Carcinoma; Radiation Exposure
MeSH Terms: conditions — Anus Neoplasms | interventions — Mn(III) meso-tetrakis(N-n-butoxyethylpyridinium-2-yl)porphyrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Concurrent Radiation Therapy, 5FU, Mitomycin and BMX-001 (Other): One arm includes all enrolled patients.
  Interventions: Drug: BMX-001

INTERVENTIONS:
Drug: BMX-001 — BMX-001 at escalating doses in combination with standard RT, 33 fractions to 59.4 Gy, plus Mitomycin at the standard dosing of 10 mg/m2 administered IV bolus at day 1 and day 29 as well as 5FU 1g/m2/d day 1-4 and 29-32.
  Other Names: MnTnBuOE-2-PyP5+; manganese butoxyethyl pyridyl porphyrin

SUMMARY:
Over 80% of anal cancers are squamous cell carcinoma (SCC). Current standard treatment for locally advanced squamous cell carcinoma of the anal canal is a combination of radiation therapy (RT) and concurrent chemotherapy. This allows for organ preservation in approximately 75% of patients. The use of concurrent radiation and chemotherapy with infusional 5-fluorouracil (5-FU) and mitomycin results in locoregional relapse rates of 20-32 and 5-year overall survival rates of 58-78%. However, while mitomycin significantly increases the rate of grade 4 toxicities, it improves local outcomes and has been considered a necessary agent in the care of anal cancer. Oxidative stress induced by radiotherapy and chemotherapy tends to protect tumor cells and promote normal tissue damage. A recently developed compound, BMX-001 (MnTnBuOE-2- PyP5+), is among the most highly potent metalloporphyrin compounds which reduce oxidative stress, thereby protecting normal tissues and augmenting tumor killing.

In this Phase 1/2 study, the investigators will conduct a safety and efficacy study of the combination of BMX-001 with standard radiation therapy and concurrent (5FU)/mitomycin in newly diagnosed Anal Squamous Cell Carcinoma (ASCC) patients. The primary Phase 1 objective is to determine the maximum tolerated dose (MTD) of BMX-001 in ASCC patients receiving RT and concurrent 5FU/mitomycin chemotherapy. Three participants will be treated at Dose Level 1 and three at Dose Level 2, then three at Dose Level 3. Dose Limiting Toxicities (DLT) experienced by any participant will be used to determine the MTD. The Phase II objective is to examine the impact of BMX-001 on the overall acute ≥ grade 3 toxicity rate of the normal tissue including rectum, bladder, and skin in combination with RT and concurrent 5FU/mitomycin in treatment of newly diagnosed ASCC patients. These will be determined by participant reports, biological materials (blood, tissue, urine) sampling and imaging. Participant health-related quality of life will be assessed by two questionnaires.

DETAILED DESCRIPTION:
Over 80% of anal cancers are squamous cell carcinoma (SCC). Current standard treatment for locally advanced squamous cell carcinoma of the anal canal is a combination of radiation therapy (RT) and concurrent chemotherapy. This allows for organ preservation in approximately 75% of patients. The use of concurrent radiation and chemotherapy with infusional 5-fluorouracil (5-FU) and mitomycin results in locoregional relapse rates of 20-32 and 5-year overall survival rates of 58-78%. However, while mitomycin significantly increases the rate of grade 4 toxicities, it improves local outcomes and has been considered a necessary agent in the care of anal cancer. Oxidative stress induced by radiotherapy and chemotherapy tends to protect tumor cells and promote normal tissue damage. A recently developed compound, BMX-001 (MnTnBuOE-2- PyP5+), is among the most highly potent metalloporphyrin compounds which reduce oxidative stress, thereby protecting normal tissues and augmenting tumor killing.

In this Phase 1/2 study, the investigators will conduct a safety and efficacy study of the combination of BMX-001 with standard radiation therapy (RT) and concurrent 5-fluorouracil (5FU)/mitomycin in newly diagnosed anal squamous cell carcinoma (ASCC) participant. A recently completed Phase 1 study using BMX-001 with concurrent chemotherapy and radiation therapy in patient with newly diagnosed high-grade gliomas (BMX-HGG-001) demonstrated no adverse effects in subcutaneous dosing up to 28 mg/subject load with half the loading dose (14 mg/subject) given biweekly for 8 weeks in 12 participants. One of three participants dosed with 42 mg/subject load with half the loading dose given biweekly for 8 weeks experienced dose-limiting toxicity (DLT) of grade 3 tachycardia and grade 3 hypotension at loading dose. These resolved with treatment within 24 hours and the participant returned to the study with no recurrence for the maintenance does. The sponsor determined that the Recommended Phase 2 Dose (RP2D) of BMX-001 is 28 mg/subject load followed by 14 mg/subject twice a week for up to eight weeks as the maximum dose that was tolerated with no adverse effects. The most common related toxicity seen in this study grade 1 injection site reaction. There is no apparent toxicity to end organ tissues or bone marrow.

For this study, after completion of Phase 1 and establishment of a RP2D for the treatment regimen in participants undergoing radiation therapy and chemotherapy, the protocol will proceed to Dose Level 3, after completion of Dose Level 1 and Dose Level 2. Up to 20 participants will be enrolled with a safety lead-in of 6 participants to confirm safety in subjects in this cohort receiving radiation therapy and 5FU/mitomycin. To evaluate the pharmacokinetics (PK) of BMX-001 in combination with current chemoradiation, blood samples will be drawn for analysis in three to six participants in enrolled in the safety lead-in. Next, the first dose of BMX-001 will be administered subcutaneously from 4 days up to 1 hour prior to the start of radiation treatment. Blood will be drawn for PK on the following days: Day 1 (before and after loading dose), Day 8, Day 22 and Day 36. Measures will be obtained at approximately the following times: -1 to 0 hour (before loading dose), 30 minutes after the drug is given, 4 hours post-dose, and 24 hours post-dose. Samples will be analyzed for BMX-001 using validated analytical methods. Skin, gastrointestinal (GI), and genitourinary (GU) symptoms will be measured on the day of screening, weekly during RT, 1 months, 4 months and 10 months after the completion of RT. Perianal skin will be assessed weekly during RT, 1 month, 4 months, and 10 months after completion of RT. Further follow up will be per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed locally advanced anal squamous cell carcinoma (including oligometastatic disease) with concurrent chemoradiation with standard Fluorouracil (5FU)/mitomycin regimen with curative intent
* Any cancer stage requiring a dose of 59.4 cGy
* 19 years of age or older
* Karnofsky Performance Status (KPS) ≥ 60%
* Hemoglobin ≥ 9.0 g/dl (a transfusion or other intervention to achieve Hgb > 9.0 g/dl is acceptable)
* Absolute neutrophil count (ANC) ≥ 1,500 /dl
* Platelets ≥ 100,000 /dl
* Serum creatinine ≤ 1.5 mg/dl, serum SGOT and bilirubin ≤ 1.5 times upper limit of normal
* Negative pregnancy test for women of child-bearing potential within 48 hours prior to first dose of BMX-001
* Use of a medically effective means of birth control until 12 months following the last study treatment for women of childbearing potential and male participants
* Positron Emission Tomography (PET)/ Computed Tomography (CT)/pelvic magnetic resonance imaging (MRI) done within 8 weeks of trial initiation

Exclusion Criteria:

* Breast-feeding
* Active infection requiring IV antibiotics within 7 days before enrollment
* Prior, unrelated malignancy requiring current active treatment, exception: cervical carcinoma in situ, basal cell or carcinoma of the skin, invasive cancers with a 5-year disease-free interval, resected cancer of the bladder, or low-grade prostate cancer (Gleason 6 or less)
* Prior history of Acantholytic squamous cell carcinoma (ASCC)
* Prior history of pelvic radiotherapy for any other type of malignancy
* Known hypersensitivity to Fluorouracil (5FU) and/or mitomycin
* Current corticosteroid use unless dose is stable or decreasing at study enrollment (anti-inflammatory properties could interrupt oxidative stress)
* Inadequately controlled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Active or history of postural hypotension and autonomic dysfunction within the past year
* Known hypersensitivity to BMX-001
* Clinically significant (active) cardiovascular disease or cerebrovascular disease, (e.g., cerebrovascular accidents ≤ 6 months prior to study enrollment, myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment
* History or evidence from physical/neurological examination of central nervous system disease (e.g. seizures) unrelated to cancer, potentially interfering with protocol treatment unless adequately controlled by medication
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis, including structural heart disease) within 6 months prior to start of study treatment
* Marked baseline prolongation of QT/QTc interval [e.g., repeated demonstration of a QTc interval >450 milliseconds (ms), CTCAE grade 1, using the specific/usual choice by clinical center for correction factor
* History of additional risk factors for Torsades de Pointes (TdP) (e.g., congestive heart failure, hypokalemia, known family history of Long QT Syndrome)
* Documented recent electrolyte disturbances (hypokalemia, hypomagnesemia, or hypocalcemia) that were clinically significant and not corrected. No additional laboratory testing is required solely for screening.
* Medical necessity for anti-arrhythmics with significant risk of QTc prolongation such as class I and class III anti-arrhythmics. These include but are not limited to amiodarone, quinidine, dofetilide, sotalol, flecainide, and lidocaine

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of BMX-001 | Within first year of the study
  Maximum tolerated dose (MTD) of BMX-001 will be determined by the highest dose level at which at least 1 out of 6 participants experienced a Dose-Limiting Toxicity (DLT).
Count of Adverse Events, Serious Adverse Events and Dose Limiting Toxicities | 10 months post-radiation therapy
  Acute grade 3 of normal tissue for adverse events (AE), serious adverse events (SAE) and dose limiting toxicities (DLT) will be recorded per Common Terminology Criteria for Adverse Events (CTCAE) 4.0.

SECONDARY OUTCOMES:
Impact of Study Treatment on Acute Rectal Bleeding | 10 months post-radiation therapy
  Acute grade 3 of normal tissue for rectal bleeding will be recorded per Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Impact of Study Treatment on Acute Rectal Pain | 10 months post-radiation therapy
  Acute grade 3 of normal tissue for rectal pain will be recorded per Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Impact of Study Treatment on Bowel Movements | 10 months post-radiation therapy
  Acute grade 3 of normal tissue for diarrhea will be recorded per Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Impact of Study Treatment on Acute Dysuria | 10 months post-radiation therapy
  Acute grade 3 of normal tissue for dysuria will be recorded per Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Impact of Study Treatment on Acute Hematuria | 10 months post-radiation therapy
  Acute grade 3 of normal tissue for hematuria will be recorded per Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Impact of Study Treatment on Acute Urinary Frequency | 10 months post-radiation therapy
  Acute grade 3 of normal tissue for urinary frequency will be recorded per Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Impact of Study Treatment on Acute Perianal Grade 3 Radiation Dermatitis | 10 months post-radiation therapy
  Acute grade 3 of normal tissue for acute perianal grade 3 radiation dermatitis will be recorded per Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Impact of Study Treatment on Late Rectal Bleeding | 10 months post-radiation therapy
  Acute grade 3 of normal tissue for late rectal bleeding per will be recorded per Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Impact of Study Treatment on Rectal Fibrosis | 10 months post-radiation therapy
  Acute grade 3 of normal tissue for rectal fibrosis will be evaluated by endoscopy.
Effect of Study Treatment on Local Control | 10 months post-radiation therapy
  The local recurrence rate will be assessed.
Effect of Study Treatment on Overall Survival | 10 months post-radiation therapy
  Overall survival (OS) rate will be determined.
Effect of Study Treatment on Locoreginal Progression-free Survival | 10 months post-radiation therapy
  Locoreginal progression-free survival rate survival (PFS) will determined.

OTHER OUTCOMES:
Effect of Study Treatment on Urine Levels of 4-hydroxynonenal | 4 months post-radiation therapy
  4-hydroxynonenal (4-HNE) will be measured in urine.
Effect of Study Treatment on Plasma Levels of 4-hydroxynonenal | 4 months post-radiation therapy
  4-hydroxynonenal (4-HNE) will be measured in plasma.
Effect of Study Treatment on Serum Level of 8-OHdG | 4 months post-radiation therapy
  8-OHdG will be measured in serum.
Effect of Study Treatment on Blood Cells Level of 8-OHdG | 4 months post-radiation therapy
  8-OHdG will be measure in blood cells.
Effect of Study Treatment on Urine Level of 8-OHdG | 4 months post-radiation therapy
  8-OHdG will be measured in urine.
Effect of Study Treatment on Urine Levels of Malondialdehyde | 4 months post-radiation therapy
  Malondialdehyde (MDA) will be measured in urine.
Effect of Study Treatment on Plasma Levels of Malondialdehyde | 4 months post-radiation therapy
  Malondialdehyde (MDA) will be measured in plasma.
Single-dose and Repeated-dose Pharmacokinetic Profiles of BMX-001 | Up to 36 days of the chemoradiation phase
  Serum drug concentration of BMX-001 will be measured after single-dose and repeated-dose BMX-001 delivery.
Effect of Study Treatment on Participant-reported Outcomes of Health-related Quality of Life | 10 months post-radiation therapy
  Participant-reported outcomes will be evaluated with the EORTC QLQ-CR29 questionnaire. This instrument consists of five functional scales, four subscales and 19 single items related to various colorectal cancer-related symptoms and functional problems. Scores can be linearly transformed to a range from 0 to 100, where higher scores generally indicate better functioning or a higher level of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Lin, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No